CLINICAL TRIAL: NCT03206658
Title: Usefulness of Spironolactone for the Prevention of Acute Kidney Injury in Critically Ill Patients With Invasive Mechanical Ventilation
Brief Title: Spironolactone on Acute Kidney Injury in Critically Ill Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: National Council of Science and Technology, Mexico (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Norma Bobadilla, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1251
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; prevention; severity; biomarker
MeSH Terms: conditions — Acute Kidney Injury | interventions — Spironolactone; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo oral capsules (Placebo Comparator): Placebo capsules equal to those in the study drug, will be administered every 24 hours for the first 5 days after entry into the critical care unit
  Interventions: Drug: Placebo oral capsule
- spironolactone (Experimental): capsules of spironolactone 25 mg equal to placebo, will be given every 24 hours for the first 5 days after entry to the critical care unit
  Interventions: Drug: Spironolactone 25 mg

INTERVENTIONS:
Drug: Spironolactone 25 mg — A dose of 25 mg of spironolactone will be administered orally or through the nasogastric /nasoenteral tube to the patients every 24 hours, at 8-9 am.
  Other Names: aldactone 25 mg
  Arms: spironolactone
Drug: Placebo oral capsule — The contents of a placebo capsule will be administered orally or through the nasogastric / nasoenteral tube to the patients every 24 hours, at 8-9 am.
  Other Names: control group
  Arms: placebo oral capsules

SUMMARY:
This study was designed to evaluate the effect of spironolactone administration in the incidence and severity of AKI in patients critically ill with invasive mechanical ventilation (IMV) in the critical care unit.

Patients in critical care unit (CCU) are the most at risk of developing AKI. In most cases a mechanism of ischemia/reperfusion has a central role in the development of AKI. Aldosterone has traditionally been recognized as a mediator that maintains water and sodium homeostasis. Nevertheless, there are enough evidence in humans and experimental models that aldosterone might mediate detrimental effects on renal function and structure in pathophysiological conditions. Indeed, several experimental studies from our laboratory have shown that mineralocorticoid receptor blockade protects the kidney against ischemia/reperfusion injury.

The aim of this study is to know:

o If mineralocorticoid receptor blockade may reduce the incidence and severity of AKI in critically patients with IMV in CCU.

You may be able to enter in this study if:

* You are at least 18 years old.
* You are male or female
* You are with IMV.
* You are in CCU.
* Your serum K is less than 4.5 mEq/L
* Your BP is >90/70 mmHg

You cannot enter this study if:

* You have CKD
* You have AKI

This study will recruit 90 patients from Instituto Nacional de Ciencias Médicas Salvador Zubiran in México City. The study will begin in April 2017. The patients will be randomized to one of 2 groups of treatment (Spironolactone 25 mg or placebo). All treatments looks identical (1 capsule), will be administered through the nasogastric tube. Neither the patients nor their doctors will be able to know or decide which group you are in. You will receive the medication during the first five days of stay in the critical care unit.

As part of this trial, the doctors will ask your permission to get a sample urine during this days. They will use the samples to do tests in the laboratory (different to routine tests) that may help them to compare renal function and biomarkers of renal injury. Your participation will end 10 days after your entry into the critical care unit. The most common side effect of spironolactone is hyperkalemia.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common multifactorial syndrome in hospitalized patients. Patients in critical care units have the highest risk of developing AKI, which is related to an increase in morbidity and doubles in-hospital mortality (10.2% vs. 25.6%) and at 90 days (16.6% vs. 33.7%).

The frequency of this condition reaches 39.3% of the critically ill patients hospitalized in the Intensive Care Units (ICU). Most cases occur early, 91% of cases occur within the first 5 days of entry. There are numerous studies in the literature investigating risk factors related to the development of AKI in critically ill patients hospitalized in critical care units. Some of those who have been associated with severe AKI and need for renal replacement therapy are: invasive mechanical ventilation, septic shock, cardiogenic shock and hepato-renal syndrome; In addition, the presence of multiple organic faults (by Sequential Organ Failure Assessment scale) is closely related to the development of AKI, and the risk seems to increase in parallel with the number of organic failures. The pathophysiological relationship between invasive mechanical ventilation and the development of AKI is well known, both for direct and indirect effects, therefore patients with invasive ventilatory support represent a special risk group.

In a recently published study evaluating the long-term prognosis of a cohort of patients who developed AKI with dialysis requirement, 62% of mortality was reported at 3.5 years, with an average survival of 8.1 to 8.9 months since the moment of dialytic requirement; almost 6% of patients in the study remained on renal replacement therapy at 3.5 years of follow-up, while 42% had micro or macroalbuminuria. (Microalbuminuria 32% and macroalbuminuria 9.9%), with a reduction in estimated glomerular flitration rate of 38 ± 29 ml/min/1.73 m2 in the 3.5 years of follow-up.

One of the major problems in the diagnosis and treatment of AKI is the difficulty in identifying it timely. From the moment of AKI occurs, the increase in the creatinine can be up to 72 h. For this reason, there is an intense search for biomarkers that allow the timely diagnosis of AKI. Several biomarkers for the early detection of AKI have been identified. These include: neutrophil gelatinase-associated lipocalin (NGAL), a protein of the lipocalin family, present in neutrophil secondary granules. Upon renal damage this protein is released from the affected epithelium early. Studies that have evaluated its usefulness as a marker of renal damage have been performed mainly in children, and its usefulness in critically ill patients has been debated. Another biomarker that has been used for the detection of renal damage is the transmembrane glycoprotein Kim-1, which releases its extracellular ectodomain by the action of proteases. Under normal conditions, Kim-1 expression is very low and increases significantly when there is tubular damage, such as occurs during AKI. A characteristic feature of this molecule is that it is expressed only in injured renal tissue. Although the induction of Kim-1 after an AKI episode is important, unfortunately this protein has not been shown to be useful as an early biomarker of AKI. Recently, our group identified a new, non-invasive, and reliable biomarker to detect AKI earlier by measuring the concentration of the 72 kilodaltons heat shock protein (HSP72). Similar to Kim-1, this protein is practically not expressed under normal conditions, but is induced in the tubular epithelium after an episode of AKI. In addition to being a highly sensitive and early biomarker, it was able to stratify different degrees of renal injury and to monitor the efficacy of a renoprotective maneuver in animals undergoing ischemia/reperfusion. In addition, we have also observed that in critically ill patients, the detection of HSP72 in urine specimens made it possible to detect AKI 48 h before diagnosis of creatinine elevation or reduction of urinary flow.

Aldosterone and kidney injury in hum There are limited number of studies aimed to evaluate the prevention of AKI with the use of any particular strategy, regard with the use of spironolactone either. However, in a study published by Dr. Brown's group in the United States aimed for decreasing the frequency of postoperative atrial fibrillation (AF) by decreasing the concentration of cytokines and inflammation that has been linked to the development of fibrillation (147 patients), ramipril (151 patients) or spironolactone 25 mg/day (147 patients) were randomly assigned to the study group. Of the secondary objectives of the study, serum K and creatinine levels were considered among other measurements. The frequency of AF in the postoperative period was similar. It should be noted that when analyzing other values such as blood pressure there were no differences between groups, despite being critically ill patients, thus the administration of these drugs did not affect AF. The need for amine use in the postoperative period was similar in the placebo group and the treatment groups. In the postoperative period, an increase in potassium levels was observed in the spironolactone group, but only in one case was necessary to suspend the treatment. The most important aspect of this study is that those patients with spironolactone or ramipril had a lower elevation of creatinine levels compared to the placebo group, which was interpreted as a prevention of renal damage independent of hemodynamic factors. Other observed results were that the group receiving spironolactone had a shorter hospital stay and a reduction in the time of invasive mechanical ventilation.

The present project has an important diagnostic potential because it will not only contribute to the early detection in the clinical practice of AKI, it will help with a new timely intervention to the patient with a novel therapy and we believe that it will also help to stratify the damage and to identify patients susceptible to developing chronic renal failure.

The AKI is a frequent complication in critically ill patients, with a reported incidence of up to 30-40% of patients entering these units. There is a directly proportional relationship between the incidence of AKI and a substantial increase in the morbidity and mortality of patients who develop it. In-hospital mortality has been reported at 35% and at 90 days up to 34%. Although AKI has a multifactorial origin, invasive mechanical ventilation (IMV) represents an independent risk factor for the development of AKI because it exerts several deleterious effects on renal perfusion and systemic inflammation. In addition, critically ill patients with IMV who will develop AKI have an increased risk of death, so the development of strategies to reduce the risk of AKI in this group of patients is of great importance.

The tools available to decrease the frequency of AKI are scarce and sometimes lack of clinical value. To date, there is no "specific" strategy, with adequate support in the literature to prevent AKI in critical ill patients.

Modifying the incidence of AKI in this group of patients will modify morbimortality related to short, medium and probably long term.

The primary involvement of aldosterone in renal damage opens a field of investigation in order to diminish or block its deleterious effects through the blockade of the mineralocorticoid receptor, in order to prevent, decrease the severity or accelerate the recovery of the AKI in these patients.

Main Hypothesis:

Administration of spironolactone will reduce significantly urinary excretion of tubular damage biomarkers such as NGAL, KIM-1 and HSP72 when compared with those of critically ill patients with invasive mechanical ventilation who will receive placebo.

Sample Size Since there is no similar study in the literature and considering a previous work of our team, in which we measured the urinary levels of HSP72 as a biomarker just at the time of diagnosis of AKI, of the 56 patients included, only 17 (30.4%) developed AKI. The mean urinary levels of HSP72 in patients who did not develop AKI were 0.27±0.16 ng/ml, whereas in those diagnosed with AKI, the mean value was 4.78±1.92 ng/ml. Considering urinary levels of HSP72 in 56 patients, the mean was 1.64 ± 2.34 ng/ml. Making a theoretical model where we consider a possible reduction of 50% of the levels of the biomarker gives us a value of 0.82 ng/ml and using the formula of sample size for independent means with the difference of means of 0.82 and equal variances with a confidence level of 95% and a power of 80%, gives us n of 45 subjects per group. Therefore, we will recruit 90 patients for this study. When 20 patients have been recruited in the study per group, an interim analysis will be performed to decide on the basis of the results if the study is continued or permanently discontinued.

variables and outcomes to be measured The analysis of the determination of the urinary concentration of NGAL, KIM-1, HSP72 and markers of oxidative stress during the evaluation period as well as the determination of the frequency of AKI will be analyzed on an exploratory basis by subgroups according to the baseline characteristics

* baseline severity of chronic diseases (Charlson comorbidity index)
* baseline severity of acute disease (APACHE II)
* previous use of spironolactone or angiotensin-converting enzyme inhibitor
* age (18-45, 45-64, 65-74, 75-90, 90)

Frequency of Measurements: for the evaluation of the primary outcome, a urinary sample per day (through the Foley catheter) during treatment periods (days 1 to 5) and surveillance Days 7 and 10 from study entry for the determination of markers of tubular damage and oxidative stress.

For the evaluation of the secondary outcome and the detection of adverse events, data will be collected for each patient since informed consent is obtained in the Selection (Day -1 to 0), treatment period (days 1 to 5), follow-up period (Days 6 to 10) and in the late evaluation visit (day 30).

Statistical analysis: the statistical analysis will be carried out by intention to treat as per protocol. Categorical variables will be shown as frequencies and proportions. The continuous variables will be analyzed with the Z of Kolmogorov-Smirnov to determine their distribution. Those with normal distribution will be shown with mean and standard deviation, while those with abnormal distribution will be presented with median and interquartile range. To compare the 2 groups Chi square for the categorical variables will be used. If it is shown that the AKI frequency is reduced, the relative risk reduction will be calculated. The numerical variables with normal distribution will be analyzed with one-way ANOVA and post hoc analysis with Bonferroni test, whereas in the case of variables with abnormal distribution, they will be analyzed with the Kruskal-Wallis test. A p less than 0.05 will be considered significant.

Potential risks: The most important adverse effects are the potential development of hypotension and hyperkalemia, however given close monitoring with multiple assessments during the day their identification will be made in a timely manner to take the necessary action. In addition, with the administration of spironolactone, general malaise and fatigue may occur, which are uncommon and mild in intensity. In cases of prolonged treatment (weeks-months) can develop gynecomastia, menstrual alterations, amenorrhea, impotence, etc.; However the likelihood of developing these alterations is very low since the exposure time will be minimal.

Safety measures for early diagnosis and prevention of risks and Early detection methods: routinely, patients with invasive mechanical ventilation in the institution are monitored closely. They usually receive monitoring of their vital signs every hour and at least a determination of creatinine, urea nitrogen in blood and electrolytes every 24 h. This will allow for the timely detection of adverse effects and suspension of study drugs if required.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Patients critically ill requiring invasive mechanical ventilation with some organic failure in addition to respiratory failure.

Organic scale failure will be categorized according to the (Sequential Organ Failure Assesment) scale and will be considered present when there is a score ≥2 in some organ / system, except renal.

* Patients with normal renal function or chronic kidney disease KDOQI 1-3
* Patients without acute renal injury according to the (acute kidney injury network) AKIN criteria.
* Normal serum K levels (less than or equal to 5 mEq / L).
* Women with (a) negative pregnancy test, (b) surgical sterilization, or (c) completed menopause.
* Systolic blood pressure> 90 mmHg and mean arterial pressure> 70 mmHg.
* Diuresis in the first 6 hrs from admission to intensive therapy> 0.5 ml / kg / hr.
* The patient will give written and signed informed consent prior to any specific study procedure. However, if a patient can not do so before, his or her legal representative the Institute may give written informed consent.

Exclusion Criteria:

* Patients with chronic kidney disease stages 4-5 of KDOQI / renal replacement therapy.
* Patients with acute kidney injury according to the AKIN criteria at the time of admission to the intensive care unit
* Patients with refractory septic shock, defined as a state of hypotension requiring administration of ≥0.25 mcg / kg / min of noradrenaline.
* Patients with known adrenal insufficiency.
* Patients with indication for the administration of angiotensin-converting enzyme (ACE) blockers or angiotensin 2 receptor antagonists.
* Known allergy to spironolactone.
* Contraindication for orally medication or placement of any probe (SNG or SNE)
* It is considered that the patient is unlikely to survive the study period (30 days) or has a disease of rapid or terminal progression.
* The patient is participating in any other clinical trial involving the administration of a research drug at the time of the presentation during the course of the study or has been treated with a research drug within 30 days prior to enrollment.
* The patient has been enrolled in this study previously.
* The patient is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
level of urinary biomarkers of AKI | at the day 0, 1, 2, 3 , 4, 5, 7 and 10 from the inclusion in the study
  determine the concentrations of NGAL, KIM-1, oxidative stress and Hsp72 in urine

CONTACTS AND LOCATIONS:
Overall Officials: Norma Bobadilla-Sandoval, PhD, Principal Investigator — INCMNSZ / IBB UNAM

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuiper JW, Groeneveld AB, Slutsky AS, Plotz FB. Mechanical ventilation and acute renal failure. Crit Care Med. 2005 Jun;33(6):1408-15. doi: 10.1097/01.ccm.0000165808.30416.ef. PMID 15942363
- [Background] Martensson J, Martling CR, Bell M. Novel biomarkers of acute kidney injury and failure: clinical applicability. Br J Anaesth. 2012 Dec;109(6):843-50. doi: 10.1093/bja/aes357. Epub 2012 Oct 9. PMID 23048068
- [Background] Han WK, Bailly V, Abichandani R, Thadhani R, Bonventre JV. Kidney Injury Molecule-1 (KIM-1): a novel biomarker for human renal proximal tubule injury. Kidney Int. 2002 Jul;62(1):237-44. doi: 10.1046/j.1523-1755.2002.00433.x. PMID 12081583
- [Background] Liangos O, Perianayagam MC, Vaidya VS, Han WK, Wald R, Tighiouart H, MacKinnon RW, Li L, Balakrishnan VS, Pereira BJ, Bonventre JV, Jaber BL. Urinary N-acetyl-beta-(D)-glucosaminidase activity and kidney injury molecule-1 level are associated with adverse outcomes in acute renal failure. J Am Soc Nephrol. 2007 Mar;18(3):904-12. doi: 10.1681/ASN.2006030221. Epub 2007 Jan 31. PMID 17267747
- [Background] Briet M, Schiffrin EL. Aldosterone: effects on the kidney and cardiovascular system. Nat Rev Nephrol. 2010 May;6(5):261-73. doi: 10.1038/nrneph.2010.30. Epub 2010 Mar 16. PMID 20234356
- [Background] Del Vecchio L, Procaccio M, Vigano S, Cusi D. Mechanisms of disease: The role of aldosterone in kidney damage and clinical benefits of its blockade. Nat Clin Pract Nephrol. 2007 Jan;3(1):42-9. doi: 10.1038/ncpneph0362. PMID 17183261
- [Background] Greene EL, Kren S, Hostetter TH. Role of aldosterone in the remnant kidney model in the rat. J Clin Invest. 1996 Aug 15;98(4):1063-8. doi: 10.1172/JCI118867. PMID 8770880
- [Background] Rocha R, Stier CT Jr, Kifor I, Ochoa-Maya MR, Rennke HG, Williams GH, Adler GK. Aldosterone: a mediator of myocardial necrosis and renal arteriopathy. Endocrinology. 2000 Oct;141(10):3871-8. doi: 10.1210/endo.141.10.7711. PMID 11014244
- [Result] Nisula S, Kaukonen KM, Vaara ST, Korhonen AM, Poukkanen M, Karlsson S, Haapio M, Inkinen O, Parviainen I, Suojaranta-Ylinen R, Laurila JJ, Tenhunen J, Reinikainen M, Ala-Kokko T, Ruokonen E, Kuitunen A, Pettila V; FINNAKI Study Group. Incidence, risk factors and 90-day mortality of patients with acute kidney injury in Finnish intensive care units: the FINNAKI study. Intensive Care Med. 2013 Mar;39(3):420-8. doi: 10.1007/s00134-012-2796-5. Epub 2013 Jan 5. PMID 23291734
- [Result] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Result] de Mendonca A, Vincent JL, Suter PM, Moreno R, Dearden NM, Antonelli M, Takala J, Sprung C, Cantraine F. Acute renal failure in the ICU: risk factors and outcome evaluated by the SOFA score. Intensive Care Med. 2000 Jul;26(7):915-21. doi: 10.1007/s001340051281. PMID 10990106
- [Result] Gallagher M, Cass A, Bellomo R, Finfer S, Gattas D, Lee J, Lo S, McGuinness S, Myburgh J, Parke R, Rajbhandari D; POST-RENAL Study Investigators and the ANZICS Clinical Trials Group. Long-term survival and dialysis dependency following acute kidney injury in intensive care: extended follow-up of a randomized controlled trial. PLoS Med. 2014 Feb 11;11(2):e1001601. doi: 10.1371/journal.pmed.1001601. eCollection 2014 Feb. PMID 24523666
- [Result] Barrera-Chimal J, Perez-Villalva R, Cortes-Gonzalez C, Ojeda-Cervantes M, Gamba G, Morales-Buenrostro LE, Bobadilla NA. Hsp72 is an early and sensitive biomarker to detect acute kidney injury. EMBO Mol Med. 2011 Jan;3(1):5-20. doi: 10.1002/emmm.201000105. Epub 2010 Dec 14. PMID 21204265
- [Result] Morales-Buenrostro LE, Salas-Nolasco OI, Barrera-Chimal J, Casas-Aparicio G, Irizar-Santana S, Perez-Villalva R, Bobadilla NA. Hsp72 is a novel biomarker to predict acute kidney injury in critically ill patients. PLoS One. 2014 Oct 14;9(10):e109407. doi: 10.1371/journal.pone.0109407. eCollection 2014. PMID 25313566
- [Result] Pretorius M, Murray KT, Yu C, Byrne JG, Billings FT 4th, Petracek MR, Greelish JP, Hoff SJ, Ball SK, Mishra V, Body SC, Brown NJ. Angiotensin-converting enzyme inhibition or mineralocorticoid receptor blockade do not affect prevalence of atrial fibrillation in patients undergoing cardiac surgery. Crit Care Med. 2012 Oct;40(10):2805-12. doi: 10.1097/CCM.0b013e31825b8be2. PMID 22824930
- [Result] Trachtman H, Weiser AC, Valderrama E, Morgado M, Palmer LS. Prevention of renal fibrosis by spironolactone in mice with complete unilateral ureteral obstruction. J Urol. 2004 Oct;172(4 Pt 2):1590-4. doi: 10.1097/01.ju.0000140445.82949.54. PMID 15371767